CLINICAL TRIAL: NCT02790177
Title: Is Hyaluronic Acid Effective in the Prevention of Post-operative Adhesion?
Brief Title: Role of Hyaluronic Acid in the Prevention of Post-operative Adhesions: a RCT
Acronym: HiB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Usman Ismat Butt, Senior Registrar, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ServicesIMSP
Record Dates: First submitted 2016-05-23; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Post Operative Adhesions
MeSH Terms: interventions — Hyaluronic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HiB (Experimental): This group will receive the compound for the reduction of adhesions
  Interventions: Drug: Hyaluronic Acid
- Normal saline (Placebo Comparator): This group will just receive normal saline to ensure blinding.
  Interventions: Drug: NORMAL SALINE

INTERVENTIONS:
Drug: Hyaluronic Acid
  Arms: HiB
Drug: NORMAL SALINE
  Arms: Normal saline

SUMMARY:
The objective of study is to determine the effect of hyaluronic acid on the formation of post-operative adhesions. It will be a randomized control trial comparing the product against normal saline.

ELIGIBILITY:
Inclusion Criteria:

- All consenting patients between the ages of 12-80, who undergo exploratory laparotomy and stoma formation

Exclusion Criteria:

Previous history of abdominal surgery History of peritoneal dialysis Patients in whom permanent stoma is formed

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
POST OPERATIVE ADHESIONS TO BE EVALUATED BY LAPAROSCOPY AT THREE MONTHS INTERVAL | 3 months

IPD SHARING:
Plan to Share IPD: No